CLINICAL TRIAL: NCT07196436
Title: Energy Recovery Ventilation and Air Cleaner Interventions to Improve Indoor Air Quality, Mold Control, and Asthma-Related Health Outcomes Among Inner-City Children and Adults in Low-Income Households
Brief Title: Asthma Intervention With Residential Ventilation and Air Cleaner (AIRVAC) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: Rebuilding Together North Texas (Unknown)
Responsible Party: Principal Investigator, Insung Kang, PhD, Assistant Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0280; HUD TXHHU0097-24 (Other Grant/Funding Number: U.S. Department of Housing and Urban Development)
Record Dates: First submitted 2025-09-02; First posted 2025-09-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Asthma Control; Pulmonary Function; Quality of Life; Stress; Sleep Quality
Keywords: Asthma; Asthma Control; Pulmonary Function; Lung Function; Quality of Life; Stress; Sleep Quality; Indoor Air Quality; Residential Ventilation; Air Cleaner; Air Filtration; Mold
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Asthma | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active ERV (Active Comparator): A group that will receive an active energy recovery ventilator for 1 year
  Interventions: Device: Energy Recovery Ventilator
- Sham ERV (Sham Comparator): A group that will receive a sham energy recovery ventilator (recirculation mode only) for 1 year
  Interventions: Device: Energy Recovery Ventilator (Sham)
- Active PAC (Active Comparator): A group that will receive an active portable air cleaner for 1 year
  Interventions: Device: Portable Air Cleaner
- Sham PAC (Sham Comparator): A group that will receive a sham portable air cleaner (HEPA filter removed) for 1 year
  Interventions: Device: Portable Air Cleaner (Sham)

INTERVENTIONS:
Device: Energy Recovery Ventilator — A mechanical ventilation system that exchanges stale indoor air with fresh outdoor air while transferring heat and moisture between the incoming and outgoing air streams
  Other Names: ERV
  Arms: Active ERV
Device: Portable Air Cleaner — A standalone home device that filters indoor air to remove particulate matter, allergens, and other pollutants
  Other Names: PAC; HEPA Air Cleaner; Residential Air Cleaner; Room Air Cleaner; Air Purifier
  Arms: Active PAC
Device: Energy Recovery Ventilator (Sham) — A home-installed ERV unit that operates in recirculation mode only, providing no fresh air exchange or heat/moisture transfer, serving as a placebo for study purposes.
  Arms: Sham ERV
Device: Portable Air Cleaner (Sham) — A portable air cleaner that appears to operate like an active unit but does not contain a HEPA filter and does not clean the air, serving as a placebo for study purposes
  Arms: Sham PAC

SUMMARY:
The primary goal of this study is to investigate the comparative long-term (i.e., 1-year) effectiveness of energy recovery ventilators (ERVs) and portable air cleaners (PACs) in reducing indoor air pollutants and mold levels and improving asthma-related health outcomes in inner-city children and adults with asthma in low-income households in the Dallas-Fort Worth (DFW) metropolitan area, TX. Secondary goals include: (1) examining associations among asthma outcomes, exposure to indoor air pollutants and mold, and housing-related factors, (2) conducting a cost-benefit analysis of ERV and PAC interventions for improving IAQ, mold control, and health outcomes, and (3) evaluating the utility of cost-effective methods and protocols for measuring IAQ and mold for indoor air pollution epidemiology studies and for providing practical information to patients and their physicians. Using a double-blind, placebo-controlled randomized controlled trial, 80 households will be assigned to receive active or placebo versions of ERVs or PACs. Environmental exposures and housing conditions will be monitored alongside comprehensive health assessments, including lung function tests and validated surveys on asthma control, quality of life, stress, and sleep quality.

DETAILED DESCRIPTION:
This study will evaluate the long-term effectiveness of energy recovery ventilators (ERVs) and portable air cleaners (PACs) in reducing indoor concentrations of air pollutants and mold, and improving health outcomes among children and adults with asthma. The study design will utilize a double-blind, placebo-controlled, 4-arm, parallel-group, randomized controlled trial with 1-year observation and 1-year intervention periods. Eligible children (n ≥ 40) and adults (n ≥ 40) with asthma from 80 households will be recruited from an applicant pool for RTNTX home retrofit programs. Participants will be randomized to receive one of four different interventions midway through the study: (1) ERV, (2) sham/placebo ERV, (3) PAC, or (4) sham/placebo PAC. All participants and field research team will be blinded to whether participants receive the active or sham/placebo intervention. ERVs will be equipped with minimum efficiency reporting value (MERV) 13 filters to capture particulate matter from incoming outdoor air, while sham/placebo ERVs will be modified to operate only in recirculation mode (no outdoor air ventilation). PACs will have high efficiency particulate air (HEPA) and carbon filters, whereas sham/placebo PACs will have the HEPA and carbon filters removed, leaving only the pre-filters. These objectives will be achieved through a combination of (i) baseline housing condition assessments for characterizing housing-related factors such as housing conditions, health and safety issues, and basic building performance, that may contribute to asthma exacerbations and affect the installation of ERVs, (ii) field measurements of indoor air pollutants (i.e., PM, VOCs, NO2, CO, and CO2) and mold levels (both air and surface samples), and (iii) comprehensive asthma outcome assessments via participant-reported health surveys for asthma control, asthma-related quality of life, stress, and sleep quality. Asthma control will be tracked monthly using the Asthma Control Test (ACT) for adults and the Childhood Asthma Control Test (C-ACT) for children. Quality of life, stress, and sleep will be assessed during home visits using validated instruments, including the 36-Item Short Form Health Survey (SF-36) and the Pediatric Quality of Life Inventory (PedsQL) for quality of life; the Perceived Stress Scale (PSS) and the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Stress measure for stress; and PROMIS Adult and Pediatric Sleep measures for sleep quality.

Results from the research are expected to identify practical and effective commercially available systems that can (1) investigate the long-term effects of different mechanisms between ERVs and PACs on IAQ, mold, and health outcomes in asthmatic children and adults; (2) provide novel data on associations among asthma outcomes, indoor air pollution and mold exposure, and housing-related factors; (3) evaluate the long-term health benefits, including reduced direct costs for asthma and estimated mortality attributable to improved IAQ and mold, versus the total costs of interventions; and (4) investigate the utility of low-cost sensors for assessing housing-related hazards and epidemiology studies, and for providing actionable information on IAQ and mold levels to patients and their physicians.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with physician-diagnosed asthma, including both adults and children aged 5-17
* Homeowners living in the DFW metropolitan area, TX

Exclusion Criteria:

* Participants living in homes with any smokers

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function (Spirometry) | Baseline; 6 months; 18 months; 24 months
  Pulmonary function will be assessed using an EasyOne Air spirometer. The primary parameters measured include Forced Expiratory Volume in 1 second (FEV₁), Forced Vital Capacity (FVC), and the FEV₁/FVC ratio.
Asthma Control Test Score | From enrollment to the end of intervention at 1 month (24 months in total)
  Asthma Control Test (ACT) for adults and Childhood Asthma Control Test (C-ACT) for children every month throughout the 2-year study.
  ACT score range: 5-25; higher scores indicate better asthma control. C-ACT score range: 0-27; higher scores indicate better asthma control.

SECONDARY OUTCOMES:
Asthma-Related Quality Of Life (Adults) | Baseline; 6 months; 18 months; 24 months
  36-Item Short Form Health Survey (SF-36) for adult participants.
  SF-36 score range: 0-100; higher scores indicate better health status.
Asthma-Related Quality Of Life (Children) | Baseline; 6 months; 18 months; 24 months
  Pediatric Quality of Life Inventory (PedsQL) for child participants.
  PedsQL score range: 0-100; higher scores indicate better quality of life.
Stress Levels | Baseline; 6 months; 18 months; 24 months
  Perceived Stress Scale (PSS) for adults and Perceived Stress Scale for Children (PSS-C) for children.
  PSS score range: 0-40; higher scores indicate worse perceived stress. PSS-C score range: 0-39; higher scores indicate worse perceived stress.
Sleep Quality | Baseline; 6 months; 18 months; 24 months
  PROMIS Sleep Disturbance Survey for both adult and child participants.
  PROMIS Sleep Disturbance score range: 20-80 (mean = 50, SD = 10); higher scores indicate worse sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Insung Kang, Ph.D., Principal Investigator — The University of Texas at Arlington
Locations (2):
- United States (2):
  - University of Texas at Arlington, Arlington, Texas
  - Rebuilding Together North Texas, Plano, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality concerns for participants and because the consent forms do not include provisions for public data sharing

REFERENCES:
- [Background] Bolen RM, Lamb JL. Guardian support of sexually abused children: a study of its predictors. Child Maltreat. 2002 Aug;7(3):265-76. doi: 10.1177/1077559502007003008. PMID 12139193
- [Background] Kang I, McCreery A, Azimi P, Gramigna A, Baca G, Hayes W, Crowder T, Scheu R, Evens A, Stephens B. Impacts of residential indoor air quality and environmental risk factors on adult asthma-related health outcomes in Chicago, IL. J Expo Sci Environ Epidemiol. 2023 May;33(3):358-367. doi: 10.1038/s41370-022-00503-z. Epub 2022 Nov 30. PMID 36450925
- [Background] Kang I, McCreery A, Azimi P, Gramigna A, Baca G, Abromitis K, Wang M, Zeng Y, Scheu R, Crowder T, Evens A, Stephens B. Indoor air quality impacts of residential mechanical ventilation system retrofits in existing homes in Chicago, IL. Sci Total Environ. 2022 Jan 15;804:150129. doi: 10.1016/j.scitotenv.2021.150129. Epub 2021 Sep 8. PMID 34798726